CLINICAL TRIAL: NCT07365345
Title: The Influence of Electrical Acupoint Stimulation at Different Frequencies on Hemodynamics During Anesthesia Induction in Patients Undergoing TAVR Surgery
Brief Title: Frequency of Electrical Acupoint Stimulation on Hypotension in TAVR Patients
Acronym: FRESH-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJH-A-20251111
Record Dates: First submitted 2025-12-30; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Transcatheter Aortic Valve Replacement (TAVR); Hemodynamic Stability; Anesthesia Induction; Electro-acupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-frequency (Experimental): The electrical stimulation is provided at a frequency of 100Hz
  Interventions: Other: electrical acupoint stimulation
- Low-frequency (Active Comparator): The electrical stimulation is provided at a frequency of 2Hz
  Interventions: Other: electrical acupoint stimulation

INTERVENTIONS:
Other: electrical acupoint stimulation — Electrical stimulation are administered at Neiguan, Jian Shi, and Baihui. The stimulation starts at 15 minutes before anesthesia induction and ends at 15 minutes after anesthesia induction.

SUMMARY:
Within 30 minutes before anesthesia, acupoint electrical stimulation at different frequencies were applied at Neiguan, Jian Shi, and Baihui. The changes in blood pressure during the anesthesia induction period were compared between the high-frequency group and the low-frequency group.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patients is 60 years or older;
* Patients who are scheduled to undergo TAVR surgery under general anesthesia;

Exclusion Criteria:

* Body mass index less than 18 kg/m2 or greater than 30 kg/m2;
* Hemodynamic instability (severe arrhythmia, decompensated heart failure);
* Hypotension after admission requiring intervention with vasoactive drugs;
* Severe liver or kidney dysfunction;
* Those who are contraindicated for electrical stimulation, including those with local skin damage, infection, or having implanted electrophysiological devices in the body.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under the curve representing the change in mean arterial pressure during the induction period relative to the baseline. | from start of induction to 15 minutes after induction
  The area under the curve (AUC) below baseline mean arterial pressure (MAP) is calculated as: ∑ (((Si - Sbaseline)+(Si-1 - Sbaseline))/2 × ΔX) where Sbaseline is the baseline MAP, Si is the MAP at the i-th minute (i = 1…15), and ΔX is the time interval between two measurements.

SECONDARY OUTCOMES:
Incidence of hypotension during the induction period | from start of induction to 15 minutes after induction
The dosage of vasoactive drugs | from start of induction to 15 minutes after induction
The incidence of major complications (cardiovascular adverse events, acute kidney injury, delirium) | from end of surgery to discharge from the hospital, at an average of 5 days
Length of hospital stay | from end of surgery to discharge from the hospital, at an average of 5 days
The rate of patients admitted to the intensive care unit (ICU) after surgery | from end of surgery to discharge from the hospital, at an average of 5 days
The rate of patients achieving the best recovery after surgery (discharged within 5 days after surgery, without major complications, no incision infection, no readmission, and survive within 30 days after surgery) | from end of surgery to 30 days after surgery
The score of the discharge quality assessment scale | at discharge from the hospital, at an average of 5 days after surgery
  Quality of Recovery, QoR-15
  15 items across 5 dimensions: physical comfort, physical independence, psychological support, emotional state, and pain.
  Each item is scored from 0 to 10. The total score ranges from 0 to 150, with a higher score representing better recovery.
  A change of 8 points or more is considered a Minimally Clinically Important Difference (MCID), meaning a meaningful improvement or decline from the patient's perspective.